CLINICAL TRIAL: NCT05780996
Title: Optimization of PVI Strategy Using QDOT Catheter. What is the Proper Energy Level for Anterior Wall of Pulmonary Veins- Intraprocedural Efficacy Comparison Between HSPD and vHPSD (The A-Q-RATE POWER Trial)
Brief Title: Efficacy of Anterior Wall PVI With QDOT Catheter - Intraprocedural Comparison Between vHPSD and HPSD Ablation.
Acronym: A-Q-RATE-POWER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Piotr Gardziejczyk, MD, MD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/2022
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; QDOT; very high power short-duration; pulmonary vein isolation; left atrial wall thickness; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very high-power short-duration (Active Comparator): A QDOT® 3.5-mm open-irrigated contact force-sensing RF ablation catheter (Biosense Webster, Inc., Irvine, CA, USA) will be used. In this group vHPSD (90W) will be performed. This power settings will be used for all ablation points.
  Interventions: Device: QMODE +
- High-power short-duration (Active Comparator): A QDOT® 3.5-mm open-irrigated contact force-sensing RF ablation catheter (Biosense Webster, Inc., Irvine, CA, USA) will be used. Ablation of the anterior aspect of the pulmonary veins will be performed with high-power short-duration (50 W) with target ablation index =550. Ablation of the posterior wall of the pulmonary veins will be performed with vHPSD (90W).
  Interventions: Device: QMODE

INTERVENTIONS:
Device: QMODE + — Atrial fibrillation radiofrequency ablation of the anterior and posterior wall with 90W (vHPSD)
  Arms: Very high-power short-duration
Device: QMODE — Atrial fibrillation radiofrequency ablation of the anterior wall with 50W (HPSD). Ablation of the posterior wall with 90 W (vHPSD)
  Arms: High-power short-duration

SUMMARY:
This study is a prospective, randomized controlled study to evaluate intraprocedural efficacy of anterior aspects of pulmonary veins insolation between very High Power Short Duration (vHPSD) and High Power Short Duration (HPSD) in patient with paroxysmal or persistent Atrial Fibrillation.

DETAILED DESCRIPTION:
This study is a dual-center, prospective, randomized controlled study to evaluate intraprocedural efficacy of anterior aspects of pulmonary veins isolation between very High Power Short Duration (vHPSD) and High Power Short Duration (HPSD) in patient with paroxysmal or persistent atrial fibrillation (AF).

Catheter ablation of atrial fibrillation with circumferential pulmonary vein isolation is an well-established method of treatment, particularly in symptomatic patients with atrial fibrillation (AF) who are ineffective or refractory to pharmacological treatment. Recurrence of pulmonary veins conduction is considered as a risk factor for future recurrence of AF. This may be partly related to the incomplete scar formation during the index ablation procedure. Constant technological progress (i.e. ablation catheters with contact force) has led to greater efficiency in obtaining complete isolation of pulmonary veins, achieving nearly 90% success rate in 12-month follow-up paroxysmal AF (CLOSE protocol). The duration of the RF application depends on the ablation index (AI), which proves that the energy has been effectively delivered to the myocardium. Currently, AI values are considered representative of RF power up to 50W. When energy above 50 W was used, the scar size was shown to be smaller than when the same AI value was used but with higher power. The safety and efficacy of novel ablation catheter QDOT (Biosense Webster, Irvine, CA, USA), that allows to deliver very high and high-power short-duration ablation, was already proven in clinical trials (QDOT FAST, Q-FFICIENCY). The benefits from using very high power short-duration ablation include: 1) shortening the duration of the procedure, 2) reducing the volume of fluids administered through the ablation electrode during RF application, which may be important in patients with heart and kidney failure, 3) reducing the frequency of collateral damages to surrounding structures of the heart (e.g. oesophagus). One of the differences related to the biophysics of RF applications between high and low energy is the range of penetration into the muscle tissue, which could impact on effectiveness of ablation. It was shown that lesions performed with vHPSD were smaller (up to 2,9 mm deep) compared to HPSD or conventional power with target AI. It is attractive for posterior wall of left atrium and can reduce peri-procedural complications. However vHPSD could be insufficient in some regions of anterior wall of the left atrium, which thickness may vary from 1 to 4 mm. Our research hypothesis is that integrated approach with different energies depending on the left atrium location is safe and lead to better efficacy than use of only vHPSD ablation in terms of first pass isolation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled for their first AF ablation procedure
2. Written informed consent
3. Paroxysmal or persistent AF
4. Age > 18

Exclusion Criteria:

1. previous ablation procedure with pulmonary vein isolation
2. lack of written informed consent
3. pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute procedural success | During ablation.
  First pass isolation of anterior wall of pulmonary veins.

SECONDARY OUTCOMES:
Number of additional RF application needed to obtain pulmonary vein isolation | during ablation
  Number of additional RF application needed to obtain pulmonary vein isolation
percentage of pulmonary vein pairs isolated with first encirclement | during ablation
  percentage of pulmonary vein pairs isolated with first encirclement
Total procedure duration | during ablation
  skin to skin procedure duration
Incidence of peri-procedural complications | during ablation
  Incidence of peri-procedural complications such as cardiac tamponade, stroke, pericardial effusion > 1 cm, TIA, vascular complications.
Fluoroscopy time | during ablation
  fluoroscopy time
Change of heart rhythm after right pulmonary veins isolation | during ablation
  Change of heart rhythm after right pulmonary veins isolation

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Gardziejczyk, MD, Principal Investigator — Department of Internal Medicine and Cardiology, Warsaw
Locations (2):
- Poland (2):
  - Centre of Postgraduate Medical Education, Department of Cardiology, Grochowski Hospital, Warsaw, Poland., Warsaw
  - Department of Internal Medicine and Cardiology with the Center for Diagnosis and Treatment of Venous Thromboembolism, Medical University of Warsaw, Warszawa, Poland, Warsaw

IPD SHARING:
Plan to Share IPD: No
We are open to collaboration but do not plan to give our data to others

REFERENCES:
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation: Executive summary. J Arrhythm. 2017 Oct;33(5):369-409. doi: 10.1016/j.joa.2017.08.001. Epub 2017 Sep 15. No abstract available. PMID 29021841
- [Background] Barkagan M, Contreras-Valdes FM, Leshem E, Buxton AE, Nakagawa H, Anter E. High-power and short-duration ablation for pulmonary vein isolation: Safety, efficacy, and long-term durability. J Cardiovasc Electrophysiol. 2018 Sep;29(9):1287-1296. doi: 10.1111/jce.13651. Epub 2018 Jun 20. PMID 29846987
- [Background] Reddy VY, Grimaldi M, De Potter T, Vijgen JM, Bulava A, Duytschaever MF, Martinek M, Natale A, Knecht S, Neuzil P, Purerfellner H. Pulmonary Vein Isolation With Very High Power, Short Duration, Temperature-Controlled Lesions: The QDOT-FAST Trial. JACC Clin Electrophysiol. 2019 Jul;5(7):778-786. doi: 10.1016/j.jacep.2019.04.009. Epub 2019 May 8. PMID 31320006
- [Background] Richard Tilz R, Sano M, Vogler J, Fink T, Saraei R, Sciacca V, Kirstein B, Phan HL, Hatahet S, Delgado Lopez L, Traub A, Eitel C, Schluter M, Kuck KH, Heeger CH. Very high-power short-duration temperature-controlled ablation versus conventional power-controlled ablation for pulmonary vein isolation: The fast and furious - AF study. Int J Cardiol Heart Vasc. 2021 Jul 26;35:100847. doi: 10.1016/j.ijcha.2021.100847. eCollection 2021 Aug. PMID 34381869
- [Background] Osorio J, Hussein AA, Delaughter MC, Monir G, Natale A, Dukkipati S, Oza S, Daoud E, Di Biase L, Mansour M, Fishel R, Valderrabano M, Ellenbogen K; Q-FFICIENCY Trial Investigators. Very High-Power Short-Duration, Temperature-Controlled Radiofrequency Ablation in Paroxysmal Atrial Fibrillation: The Prospective Multicenter Q-FFICIENCY Trial. JACC Clin Electrophysiol. 2023 Apr;9(4):468-480. doi: 10.1016/j.jacep.2022.10.019. Epub 2023 Jan 18. PMID 36752484
- [Background] Natale A, Reddy VY, Monir G, Wilber DJ, Lindsay BD, McElderry HT, Kantipudi C, Mansour MC, Melby DP, Packer DL, Nakagawa H, Zhang B, Stagg RB, Boo LM, Marchlinski FE. Paroxysmal AF catheter ablation with a contact force sensing catheter: results of the prospective, multicenter SMART-AF trial. J Am Coll Cardiol. 2014 Aug 19;64(7):647-56. doi: 10.1016/j.jacc.2014.04.072. PMID 25125294
- [Background] Yavin HD, Leshem E, Shapira-Daniels A, Sroubek J, Barkagan M, Haffajee CI, Cooper JM, Anter E. Impact of High-Power Short-Duration Radiofrequency Ablation on Long-Term Lesion Durability for Atrial Fibrillation Ablation. JACC Clin Electrophysiol. 2020 Aug;6(8):973-985. doi: 10.1016/j.jacep.2020.04.023. PMID 32819533
- [Background] Leshem E, Zilberman I, Tschabrunn CM, Barkagan M, Contreras-Valdes FM, Govari A, Anter E. High-Power and Short-Duration Ablation for Pulmonary Vein Isolation: Biophysical Characterization. JACC Clin Electrophysiol. 2018 Apr;4(4):467-479. doi: 10.1016/j.jacep.2017.11.018. Epub 2018 Feb 2. PMID 30067486
- [Background] Lozano-Granero C, Franco E, Matia-Frances R, Hernandez-Madrid A, Sanchez-Perez I, Zamorano JL, Moreno J. Characterization of high-power and very-high-power short-duration radiofrequency lesions performed with a new-generation catheter and a temperature-control ablation mode. J Cardiovasc Electrophysiol. 2022 Dec;33(12):2528-2537. doi: 10.1111/jce.15676. Epub 2022 Sep 24. PMID 36116038